CLINICAL TRIAL: NCT00075504
Title: A Phase II Study of Triapine in Combination With Gemcitabine in Adenocarcinoma of the Biliary Ducts and Gall Bladder
Brief Title: Triapine and Gemcitabine Hydrochloride in Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03030; 6254 (Other: CTEP); U01CA062505 (NIH); N01CM62204 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2013-05

CONDITIONS: Stage II Gallbladder Cancer; Stage IIIA Gallbladder Cancer; Stage IIIB Gallbladder Cancer; Stage IVA Gallbladder Cancer; Stage IVB Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- triapine, gemcitabine (Experimental): Triapine IV over 4 hours followed by gemcitabine IV over 30 minutes on days 1, 8, and 15, repeat every 28 days
  Interventions: Drug: triapine; Drug: gemcitabine

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Drug: gemcitabine — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; Gemzar

SUMMARY:
This phase II trial is studying how well giving 3-AP together with gemcitabine works in treating patients with unresectable or metastatic bile duct or gallbladder cancer. Drugs used in chemotherapy, such as 3-AP and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. 3-AP may help gemcitabine kill more cancer cells by making them more sensitive to the drug.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the objective response rates for the combination of triapine and gemcitabine in patients with primary tumors of the biliary ducts and gall bladder.

II. To assess the toxicities and recovery from toxicities for patients with biliary duct and gall bladder tumors treated with the combination of triapine and gemcitabine.

III. To determine the survival and progression free survival of patients with biliary and gall bladder tumors treated with the combination of triapine and gemcitabine.

OUTLINE: This is a non-randomized, multicenter study. Patients are stratified according to bilirubin levels (normal vs abnormal).

Patients receive 3-AP (Triapine) IV over 4 hours followed by gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 1 additional course beyond CR.

Patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the biliary ducts that is unresectable and/or metastatic; this can include unresectable or metastatic carcinomas of the Ampulla of Vater. In addition, unresectable or metastatic gall bladder carcinoma will be allowed
* Measurable disease
* No prior chemotherapy
* Life expectancy of greater than 3 months
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Creatinine within normal institutional limits
* Patients may have mildly abnormal liver function defined as a total bilirubin > ULN and =< 3x the institutional upper limits of normal (includes CTCAE v.3 grades 1-2 hyperbilirubinemia)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Triapine or gemcitabine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Uncontrolled pulmonary disease including asthma, chronic bronchitis and COPD or with requirements for chronic oxygen use
* Pregnant or lactating women
* HIV infection
* Patients with G6PD deficiency will be excluded in view of the potential for methemoglobinemia
* Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Ocean, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Ocean AJ, Christos P, Sparano JA, Matulich D, Kaubish A, Siegel A, Sung M, Ward MM, Hamel N, Espinoza-Delgado I, Yen Y, Lane ME. Phase II trial of the ribonucleotide reductase inhibitor 3-aminopyridine-2-carboxaldehydethiosemicarbazone plus gemcitabine in patients with advanced biliary tract cancer. Cancer Chemother Pharmacol. 2011 Aug;68(2):379-88. doi: 10.1007/s00280-010-1481-z. Epub 2010 Oct 28. PMID 20981545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 patients were enrolled from 7 institutions between December 2003 and August 2007
Pre-assignment Details: A total of 2 patients did not receive treatment
Groups:
- Stratum A Normal Liver Function Triapine, Gemcitabine; Stratum B Abnormal Liver Function Triapine, Gemcitabine: Triapine IV over 4 hours followed by gemcitabine IV over 30 minutes on days 1, 8, and 15, repeat every 28 days
  triapine: Given IV
  gemcitabine: Given IV
Period: Overall Study
Arm/Group | Stratum A Normal Liver Function Triapine, Gemcitabine | Stratum B Abnormal Liver Function Triapine, Gemcitabine
Started | 23 | 10
Completed | 14 | 3
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Stratum A Normal Liver Triapine, Gemcitabine; Stratum B Abnormal Liver Triapine, Gemcitabine: Triapine IV over 4 hours followed by gemcitabine IV over 30 minutes on days 1, 8, and 15, repeat every 28 days
  triapine: Given IV
  gemcitabine: Given IV
- Total: Total of all reporting groups
Arm/Group | Stratum A Normal Liver Triapine, Gemcitabine | Stratum B Abnormal Liver Triapine, Gemcitabine | Total
Number analyzed (Participants) | 23 | 10 | 33
Age, Continuous [Median (Full Range); unit: years] | 57 [35 to 85] | 67.5 [55 to 75] | 62.3 [35 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 12 | 4 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 10 | 30
  Black | 1 | 0 | 1
  Asian | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate According to RECIST Criteria
Description: Tumor response was assessed every eight weeks by CT scan using RECIST (Response Evaluation Criteria in Solid Tumors) criteria. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disapperance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall response (OR) = CR+PR.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Stratum A Normal Liver Function Triapine, Gemcitabine | Stratum B Abnormal Liver Function Triapine, Gemcitabine
Number analyzed (Participants) | 23 | 10
participants | 3 | 0

2. Secondary Outcome: Progression Free Survival
Description: PFS will be measured from the time of the patient's initial best response (PR or CR) until documented progression.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum A Normal Liver Function Triapine, Gemcitabine | Stratum B Abnormal Liver Function Triapine, Gemcitabine
Number analyzed (Participants) | 23 | 10
months | 3.7 [2.7 to 5.8] | 3.6 [1.9 to 11.6]

3. Secondary Outcome: Overall Survival
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum A Normal Liver Function Triapine, Gemcitabine | Stratum B Abnormal Liver Function Triapine, Gemcitabine
Number analyzed (Participants) | 23 | 10
months | 10.3 [5.9 to NA] — For stratum A the upper limit in the 95% CI for overall survival was not reached. | 3.6 [2.1 to 26.2]

ADVERSE EVENTS:
Arm/Group | Stratum A Normal Liver Function Triapine, Gemcitabine | Stratum B Abnormal Liver Function Triapine, Gemcitabine
Serious Adverse Events (participants affected / at risk) | 21/23 | 10/10
Other Adverse Events (participants affected / at risk) | 22/23 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A Normal Liver Function Triapine, Gemcitabine (N=23) | Stratum B Abnormal Liver Function Triapine, Gemcitabine (N=10)
Infection with normal ANC or Grade 1 or 2 Neutrophils: Blood (Infections and infestations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 3 (3)
Neutrophil count decreased (Investigations) | 10 (10) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 5 (5) | 4 (4)
Infection (Infections and infestations) | 7 (7) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A Normal Liver Function Triapine, Gemcitabine (N=23) | Stratum B Abnormal Liver Function Triapine, Gemcitabine (N=10)
Platelet count decreased (Investigations) | 11 (23) | 4 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Lymphocyte count decreased (Investigations) | 13 (13) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 19 (19) | 6 (6)
Alkaline phosphatase increase (Investigations) | 6 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Fatigue (General disorders) | 11 (11) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less